CLINICAL TRIAL: NCT04343937
Title: Retrolaminar Block for Postoperative Analgesia in Lumbar Herniectomy Surgery
Status: Completed | Type: Observational
Sponsor: Erzincan University (Other)
Responsible Party: Principal Investigator, Nurcan Kutluer Karaca, Assistant Professor, Erzincan University
Other Study IDs: Erzincan Binali Y. University
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Postoperative Pain
Keywords: Retrolaminar block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrolaminar block: Retrolaminar block for postoperative pain managment in patients undergoing lumbar herniectomy under general anesthesia
  Interventions: Procedure: retrolaminar block
- İntravenous analgesia: İntravenous analgesia for postoperative pain managment in patients undergoing lumbar herniectomy under general anesthesia

INTERVENTIONS:
Procedure: retrolaminar block — local anesthetic injection on the between the lamina of the vertebra and the paraspinous muscle
  Groups: Retrolaminar block

SUMMARY:
This retrospective study included 30 patients scheduled for lumbar herniectomy under general anesthesia. The patients were randomized to receive either retrolaminar block or intravenous analgesia treatment.Numeric Pain Rating Scale (NPRS) was used to measure the pain intensity of patients in postoperative period. Postoperative analgesic requirements were recorded to asses effectiveness of regional anesthesia.Opiod and NSAİD as rescue medication were recorded postoperatively.

DETAILED DESCRIPTION:
This retrospective study included 30 patients scheduled for lumbar herniectomy under general anesthesia. The patients were randomized to receive either RLB or intravenous analgesia treatment. All patients were routinely monitored and their heart rate, blood pressure and pulse oxymetry recorded during the anesthesia. Numeric Pain Rating Scale (NPRS) scores evaluated at 2, 8, 12, 24 and 48 h after the surgery. Opiod and NSAİD as rescue medication were recorded postoperatively

ELIGIBILITY:
Inclusion Criteria:

* patients accepted to part in the study

Exclusion Criteria:

* patients not accepted to part in the study
* allergic reaction to local anesthetics drugs
* lumbar herniectomy of more than two levels

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients underwent retrolaminar block
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
postoperative pain: Numeric Pain Rating Scale | at the second hour after the surgery
  Pain intensity of patients with the Numeric Pain Rating Scale after surgery. The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. Zero means the lowest score and no pain.Ten means the highest score and worst pain experienced.
postoperative pain: Numeric Pain Rating Scale | at the eighth hour after the surgery
  pain intensity of patients with the Numeric Pain Rating Scale after surgery. Pain intensity of patients with the Numeric Pain Rating Scale after surgery. The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. Zero means the lowest score and no pain.Ten means the highest score and worst pain experienced.
postoperative pain: Numeric Pain Rating Scale | at the twelfth hour after the surgery
  pain intensity of patients with the Numeric Pain Rating Scale after surgery. Pain intensity of patients with the Numeric Pain Rating Scale after surgery. The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. Zero means the lowest score and no pain.Ten means the highest score and worst pain experienced.
postoperative pain: Numeric Pain Rating Scale | at the twenty forth hour after the surgery
  pain intensity of patients with the Numeric Pain Rating Scale after surgery. Pain intensity of patients with the Numeric Pain Rating Scale after surgery. The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. Zero means the lowest score and no pain.Ten means the highest score and worst pain experienced.
postoperative pain: Numeric Pain Rating Scale | at the forty-eighth hour after the surgery
  pain intensity of patients with the Numeric Pain Rating Scale after surgery. Pain intensity of patients with the Numeric Pain Rating Scale after surgery. The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. Zero means the lowest score and no pain.Ten means the highest score and worst pain experienced.

SECONDARY OUTCOMES:
postoperative analgesic requirements | at the second hour after the surgery
  Opiod and Nonsteroidal Anti-inflammatory Drugs as rescue medication recorded postoperatively.
postoperative analgesic requirements | at the eighth hour after the surgery
  Opiod and Nonsteroidal Anti-inflammatory Drugs as rescue medication recorded postoperatively.
postoperative analgesic requirements | at the twelfth hour after the surgery
  Opiod and Nonsteroidal Anti-inflammatory Drugs as rescue medication recorded postoperatively.
postoperative analgesic requirements | at the twenty forth hour after the surgery
  Opiod and Nonsteroidal Anti-inflammatory Drugs as rescue medication recorded postoperatively.
postoperative analgesic requirements | at the forty-eighth hour after the surgery
  Opiod and Nonsteroidal Anti-inflammatory Drugs as rescue medication recorded postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Nurcan Kutluer Karaca, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No